CLINICAL TRIAL: NCT01027351
Title: A Phase 2, Open-Label, Single-Center, Extension Study Evaluating Antibody Persistence Compared to Naïve Children and Safety, Tolerability and Immunogenicity of Booster Doses of Novartis rMenB±OMV NZ Vaccine in Healthy UK Children Who Previously Received One or Four Doses of the Novartis Vaccine as Infants in Study V72P6
Brief Title: Extension Study Evaluating Antibody Persistence and Safety, Tolerability and Immunogenicity of Booster Doses of Novartis rMenB±OMV NZ Vaccine in Healthy UK Children Who Previously Received One or Four Doses of the Same Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72P6E1; EUDRACT 2009-013054-33
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Meningococcal Disease
Keywords: Children; Pre-school; Meningococcal disease; Prevention; Vaccination
MeSH Terms: conditions — Meningococcal Infections

ARMS (6):
- 5rMenB (Experimental): Subjects who had received four doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine, without Outer Membrane Vesicles (OMV) (at 2,4,6 and 12 months of age) in the parent study were administered a fifth dose of the same vaccine, at 40 months of age in the present study.
  Interventions: Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine, without Outer Membrane Vesicles (OMV)
- 5rMenB+OMV NZ (Experimental): Subjects who had received four doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine (at 2,4,6 and 12 months of age) in the parent study were administered a fifth dose of the same vaccine, at 40 months of age in the present study.
  Interventions: Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine.
- 3rMenB (Experimental): Subjects who had previously received one dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine without OMV (at 12 months of age) were administered two doses of the same vaccine, at 40 and 42 months of age in the present study.
  Interventions: Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine, without Outer Membrane Vesicles (OMV)
- 3rMenB+OMV NZ (Experimental): Subjects who had previously received one dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine (at 12 months of age) were administered two doses of the same vaccine, at 40 and 42 months of age in the present study.
  Interventions: Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine.
- Naive_4042 (Experimental): Vaccine-naive subjects who received two catch-up doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine at 40 and 42 months of age in the present study.
  Interventions: Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine.
- Naive_6062 (Experimental): Vaccine-naive subjects who received two catch-up doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine at 60 and 62 months of age in the present study.
  Interventions: Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine.

INTERVENTIONS:
Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine. — Subjects received either one or two booster doses of the same vaccine they had received in the parent trial (rMenB+OMV NZ) or two catch-up doses.
  Arms: 3rMenB+OMV NZ; 5rMenB+OMV NZ; Naive_4042; Naive_6062
Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine, without Outer Membrane Vesicles (OMV) — Subjects received either one or two booster doses of the same vaccine they had received in the parent trial (rMenB).
  Arms: 3rMenB; 5rMenB

SUMMARY:
The proposed study V72P6E1 is an Extension Study of V72P6 (NCT00381615). The objectives of this extension study will be to explore antibody persistence at approximately 40 months of age and to evaluate the safety, tolerability and immunogenicity of booster doses of rMenB±OMV NZ administered to subjects at approximately 40 months of age. Antibody persistence will be subsequently measured at 18-20 months after these booster doses when the subjects are 60 months of age. Two groups of naïve subjects, aged approximately 40 and 60 months, will be recruited in the study to serve as a baseline comparator for assessing antibody persistence at these ages. These subjects will receive a two-dose catch-up regimen with rMenB+OMV NZ. Subjects who are enrolled at 40 months of age are offered DTaP/IPV and MMR vaccinations, if they have not already received these vaccines prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 40 to 44-months-old children, who participated and completed the study V72P6 (NCT00381615; follow-on subjects)
* Healthy 40 to 44-months or 60 to 62-months-old children (naïve subjects)

Exclusion Criteria:

* Previous ascertained or suspected disease caused by N. meningitidis
* History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component
* Any serious chronic or progressive disease
* Known or suspected impairment/alteration of the immune system
* Receipt of, or intent to immunize with another vaccine, within 30 days prior and after vaccination with the investigational vaccines (within 14 days for licensed flu vaccines)

Ages: 40 Months to 62 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] McQuaid F, Snape MD, John TM, Kelly S, Robinson H, Yu LM, Toneatto D, D'Agostino D, Dull PM, Pollard AJ. Persistence of specific bactericidal antibodies at 5 years of age after vaccination against serogroup B meningococcus in infancy and at 40 months. CMAJ. 2015 Apr 21;187(7):E215-E223. doi: 10.1503/cmaj.141200. Epub 2015 Mar 23. PMID 25802309
- [Derived] Snape MD, Saroey P, John TM, Robinson H, Kelly S, Gossger N, Yu LM, Wang H, Toneatto D, Dull PM, Pollard AJ. Persistence of bactericidal antibodies following early infant vaccination with a serogroup B meningococcal vaccine and immunogenicity of a preschool booster dose. CMAJ. 2013 Oct 15;185(15):E715-24. doi: 10.1503/cmaj.130257. Epub 2013 Sep 23. PMID 24062178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 1 center in the United Kingdom.
Pre-assignment Details: All subjects were included in the trial.
Groups:
- 5rMenB: Subjects who had received four doses of rMenB vaccine (at 2,4,6 and 12 months of age) in the parent study were administered a fifth dose of rMenB vaccine, at 40 months of age in the present study.
- 5rMenB+OMV NZ: Subjects who had received four doses of rMenB +OMV NZ vaccine (at 2,4,6 and 12 months of age) in the parent study were administered a fifth dose of rMenB +OMV NZ vaccine, at 40 months of age in the present study.
- 3rMenB: Subjects who had previously received one dose of rMenB vaccine (at 12 months of age) were administered two doses of rMenB vaccine, at 40 and 42 months of age in the present study.
- 3rMenB+OMV NZ: Subjects who had previously received one dose of rMenB +OMV NZ vaccine (at 12 months of age) were administered two doses of rMenB +OMV NZ vaccine, at 40 and 42 months of age in the present study.
- Naive_4042: Vaccine-naive subjects who received two catch -up doses of rMenB+OMV NZ vaccine at 40 and 42 months of age in the present study.
- Naive_6062: Vaccine-naive subjects who received two catch-up doses of rMenB+OMV NZ vaccine at 60 and 62 months of age in the present study
Period: Overall Study
Arm/Group | 5rMenB | 5rMenB+OMV NZ | 3rMenB | 3rMenB+OMV NZ | Naive_4042 | Naive_6062
Started | 29 | 19 | 14 | 8 | 43 | 50
Completed | 26 | 18 | 13 | 6 | 32 | 45
Not Completed | 3 | 1 | 1 | 2 | 11 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 3 | 5
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 6 | 0
Not completed — Inappropriate enrollment | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was done on the all enrolled set.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5rMenB | 5rMenB+OMV NZ | 3rMenB | 3rMenB+OMV NZ | Naive_4042 | Naive_6062 | Total
Number analyzed (Participants) | 29 | 19 | 14 | 8 | 43 | 50 | 163
Age, Continuous [Mean (Standard Deviation); unit: months] | 41.4 (1.5) | 41.8 (1.4) | 41.4 (1.5) | 40.4 (0.7) | 41.8 (1.7) | 61.3 (0.9) | 47.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 5 | 3 | 23 | 27 | 84
  Male | 12 | 10 | 9 | 5 | 20 | 23 | 79
Region of Enrollment [Number; unit: Subjects]
  United Kingdom | 29 | 19 | 14 | 8 | 43 | 50 | 163

OUTCOME MEASURES:

1. Primary Outcome: Persistence of Geometric Mean Antibody Titers in Children (Who Previously Received 4 Doses of Men B Vaccine), at 40 Months of Age.
Description: Persistence of geometric mean titers (GMTs) against N.meningitidis B strains in children (at 40 months of age) who had previously received four doses of either rMenB or rMen+OMV NZ vaccines in parent study, are compared with the GMTs in vaccine-naïve children.
Time Frame: 28 months after last vaccination; Baseline for Naïve
Population: The analysis was done on the Modified- Intended to treat (MITT), 40 months of age, antibody persistence population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 5rMenB | 5rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 29 | 17 | 40
Titers
  H 44/76 strain | 3.24 [2.33 to 4.52] | 5.34 [3.47 to 8.23] | 4.25 [3.22 to 5.6]
  5/99 strain (N=28, 17, 40) | 5.11 [2.33 to 11] | 28 [10 to 77] | 1.11 [0.9 to 1.36]
  NZ 98/254 strain | 1.09 [0.79 to 1.51] | 2.77 [1.81 to 4.23] | 1 [1 to 1]
  M10713 strain (N=28, 15, 40) | 9.15 [5.01 to 17] | 5.34 [2.35 to 12] | 8.75 [5.22 to 15]

2. Primary Outcome: Percentage of Subjects (Who Previously Received 4 Doses of Men B Vaccine) With Persisting Human Complement Serum Bactericidal Antibody Titers ≥ 1:4 and ≥1:8 at 40 Months of Age.
Description: The percentages of subjects with persisting human serum bactericidal antibodies (hSBA) titers ≥ 1:4 and ≥ 1:8, against N.meningitidis B strains at 40 months of age; who had previously received four doses of either rMenB or rMen+OMV NZ vaccines in parent study are reported.
  The serum bactericidal antibodies directed against serogroup B meningococci, are measured by human complement Serum Bactericidal Assay (hSBA).
Time Frame: 28 months after last vaccination; baseline for naïve
Population: The analysis was done on the MITT , 40 months of age, antibody persistence population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 5rMenB | 5rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 29 | 17 | 40
Percentages of subjects
  hSBA ≥1:4 (H44/76 strain) | 45 [26 to 64] | 65 [38 to 86] | 63 [46 to 77]
  hSBA≥1:4 (5/99 strain; N=28, 17, 40) | 43 [24 to 63] | 76 [50 to 93] | 3 [0.063 to 13]
  hSBA≥1:4 (NZ 98/254 strain) | 3 [0.087 to 18] | 41 [18 to 67] | 0 [0 to 9]
  hSBA≥1:4 (M10713 strain; N=28, 15, 40) | 68 [48 to 84] | 67 [38 to 88] | 68 [51 to 81]
  hSBA ≥1:8 (H44/76 strain) | 14 [4 to 32] | 35 [14 to 62] | 30 [17 to 47]
  hSBA≥1:8 (5/99 strain; N=28, 17, 40) | 43 [24 to 63] | 76 [50 to 93] | 3 [0.063 to 13]
  hSBA≥1:8 (NZ 98/254 strain) | 0 [0 to 12] | 24 [7 to 50] | 0 [0 to 9]
  hSBA≥1:8 (M10713 strain; N=28, 15, 40) | 61 [41 to 78] | 40 [16 to 68] | 45 [29 to 62]

3. Primary Outcome: Number of Subjects Reporting Solicited Adverse Events After a Receiving One or Two Booster Doses of rMen B or rMenB+OMV NZ Vaccine at 40 Months of Age.
Description: The safety and tolerability of one or two booster doses of rMen B or rMenB+OMV NZ vaccine administered at 40 months of age in children who had previously received one or four doses of the same vaccine as infants in parent study is assessed in terms of number of subjects with solicited local and systemic reactions following vaccination.
Time Frame: Day 1-7 after booster vaccination
Population: Analysis was done on the safety population i.e all subjects who received at least one Men B vaccination and provided post-baseline safety data.
Measure: Number; unit: participants
Arm/Group | 5rMenB | 5rMenB+OMV NZ | 3rMenB | 3rMenB+OMV NZ
Number analyzed (Participants) | 29 | 19 | 14 | 8
participants
  Local | 28 | 19 | 14 | 8
  Injection-site pain | 17 | 14 | 8 | 8
  Injection-site erythema | 28 | 19 | 14 | 8
  Injection-site swelling | 13 | 5 | 9 | 4
  Injection-site induration | 14 | 9 | 8 | 6
  Systemic | 19 | 13 | 11 | 8
  Changes in eating habits | 5 | 10 | 5 | 4
  Sleepiness | 13 | 12 | 8 | 6
  Vomiting | 1 | 3 | 3 | 0
  Diarrhea | 3 | 1 | 3 | 1
  Irritability | 14 | 10 | 9 | 8
  Headache | 1 | 0 | 2 | 1
  Arthralgia | 0 | 6 | 4 | 4
  Rash | 3 | 0 | 2 | 1
  Fever (≥38°C) | 1 | 1 | 4 | 0
  Other | 10 | 12 | 5 | 7
  Antipyretic preventive medication used | 10 | 12 | 3 | 7
  Antipyretic treatment medication used | 1 | 2 | 4 | 0
  Medically attended fever | 0 | 0 | 1 | 0

4. Secondary Outcome: Persistence of Geometric Mean Antibody Titers in Children (Who Previously Received One Dose of Men B Vaccine), at 40 Months of Age.
Description: Persisting GMTs against N.meningitidis B strains in children (at 40 months of age) who had previously received one dose of either rMenB or rMen+OMV NZ vaccines in parent study, are compared with the GMTs in vaccine-naïve children.
Time Frame: 28 months after vaccination; Baseline for Naïve
Population: The analysis was done on the MITT, 40 months of age, antibody persistence population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- 3rMenB: Subjects who had previously received one dose of rMenB vaccine (at 12 months of age) in the parent study, were administered two doses of rMenB vaccine, at 40 and 42 months of age in the present study.
- 3rMenB+OMV NZ: Subjects who had previously received one dose of rMenB +OMV NZ vaccine (at 12 months of age) in the parent study, were administered two doses of rMenB +OMV NZ vaccine, at 40 and 42 months of age in the present study.
Arm/Group | 3rMenB | 3rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 14 | 8 | 40
Titers
  H44/76 strain | 3.59 [1.8 to 7.15] | 3.47 [1.39 to 8.64] | 4.25 [3.22 to 5.6]
  5/99 strain | 9.57 [3.88 to 24] | 1 [0.3 to 3.3] | 1.11 [0.9 to 1.36]
  NZ 98/254 strain | 1.23 [0.96 to 1.57] | 1 [0.72 to 1.38] | 1 [1 to 1]
  M10713 strain (N=13, 8, 40) | 3.26 [1.49 to 7.11] | 3 [1.11 to 8.11] | 8.75 [5.22 to 15]

5. Secondary Outcome: Percentage of Subjects (Who Had Previously Received One Dose of Men B Vaccine) With Persisting Serum Bactericidal Antibody Titers ≥ 1:4 and ≥1:8, at 40 Months of Age.
Description: The percentages of subjects with persisting hSBA titers ≥ 1:4 and ≥1:8, against N.meningitidis B strains at 40 months of age; who had previously received one dose of either rMenB or rMen+OMV NZ vaccines in parent study are reported.
Time Frame: 28 months after vaccination; baseline for naïve
Population: The analysis was done on the MITT, 40 months of age, antibody persistence population.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 3rMenB | 3rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 14 | 8 | 40
percentage of subjects
  hSBA ≥1:4 (H44/76 strain) | 57 [29 to 82] | 38 [9 to 76] | 63 [46 to 77]
  hSBA≥1:4 (5/99 strain) | 57 [29 to 82] | 0 [0 to 37] | 3 [0.063 to 13]
  hSBA≥1:4 (NZ 98/254 strain) | 7 [0 to 34] | 0 [0 to 37] | 0 [0 to 9]
  hSBA≥1:4 (M10713 strain; N=13, 8, 40) | 54 [25 to 81] | 25 [3 to 65] | 68 [51 to 81]
  hSBA ≥1:8 (H44/76 strain) | 7 [0 to 34] | 13 [0 to 53] | 30 [17 to 47]
  hSBA≥1:8 (5/99 strain) | 43 [18 to 71] | 0 [0 to 37] | 3 [0.063 to 13]
  hSBA≥1:8 (NZ 98/254 strain) | 0 [0 to 23] | 0 [0 to 37] | 0 [0 to 9]
  hSBA≥1:8 (M10713 strain; N=13, 8, 40) | 15 [2 to 45] | 13 [0 to 53] | 45 [29 to 62]

6. Secondary Outcome: Geometric Mean Antibody Titers in Children (Who Previously Received 4 Doses of Men B Vaccine), After Receiving a Booster Dose of rMenB or rMenB+OMV NZ Vaccine at 40 Months of Age.
Description: The GMTs against N.meningitidis B strains in children (who had previously received four doses MenB vaccine in parent study) after a single booster dose of rMenB or rMenB+OMV NZ vaccine given at 40 months of age, are compared with the antibody titers following one catch-up dose rMenB+OMV NZ vaccine given at 40 months to vaccine-naive subjects.
Time Frame: 1 month post- booster/ dose 1 for Naïve
Population: The analysis was done on the MITT population, booster response.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 5rMenB | 5rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 29 | 19 | 38
Titers
  H44/76 strain | 99 [67 to 145] | 89 [56 to 141] | 12 [7.96 to 19]
  5/99 strain (N=28, 18, 38) | 778 [448 to 1349] | 1708 [859 to 3396] | 22 [12 to 40]
  NZ 98/254 strain | 1.64 [0.95 to 2.85] | 47 [24 to 91] | 7.73 [4.62 to 13]
  M10713 strain (N=28, 18, 38) | 38 [24 to 59] | 39 [22 to 67] | 11 [6.7 to 19]

7. Secondary Outcome: Percentage of Subjects (Who Previously Received 4 Doses of Men B Vaccine) With Serum Bactericidal Antibody Titers ≥ 1:4 and ≥1:8 After Receiving a Booster Dose of Either rMenB or rMenB+OMV NZ Vaccine at 40 Months of Age.
Description: The percentages of subjects (who had previously received four doses MenB vaccine in parent study) with hSBA titers ≥ 1:4 and ≥ 1:8, against N.meningitidis B strains after receiving a single booster dose of either rMenB or rMen+OMV NZ vaccines at 40 months of age are compared with hSBA responses following one catch-up dose of rMenB+OMV NZ vaccine given at 40 months in vaccine-naive subjects .
Time Frame: 1 month post- booster/ dose 1 for Naïve
Population: The analysis was done on the MITT population, booster response.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 5rMenB | 5rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 28 | 19 | 38
Percentage of subjects
  hSBA ≥1:4 (H44/76 strain) | 100 [88 to 100] | 100 [82 to 100] | 89 [75 to 97]
  hSBA≥1:4 (5/99 strain; N=28, 18, 38) | 100 [88 to 100] | 100 [81 to 100] | 76 [60 to 89]
  hSBA≥1:4 (NZ 98/254 strain) | 14 [4 to 33] | 89 [67 to 99] | 66 [49 to 80]
  hSBA≥1:4 (M10713 strain; N=28, 18, 38) | 96 [82 to 100] | 94 [73 to 100] | 76 [60 to 89]
  hSBA ≥1:8 ( H44/76 strain) | 96 [82 to 100] | 100 [82 to 100] | 63 [46 to 78]
  hSBA≥1:8 (5/99 strain; N=28, 18, 38) | 100 [88 to 100] | 100 [81 to 100] | 71 [54 to 85]
  hSBA≥1:8 (NZ 98/254 strain) | 11 [2 to 28] | 89 [67 to 99] | 58 [41 to 74]
  hSBA≥1:8 (M10713 strain; N=28, 18, 38) | 89 [72 to 98] | 94 [73 to 100] | 61 [43 to 76]

8. Secondary Outcome: Percentage of Subjects (Who Previously Received 4 Doses of Men B Vaccine) With 4-fold Increase in Serum Bactericidal Antibody Titers After Receiving a Booster Dose of Either rMenB or rMenB+OMV NZ Vaccine at 40 Months of Age.
Description: The percentages of subjects (who had previously received four doses MenB vaccine in parent study) showing a 4-fold increase in hSBA titers over baseline against N.meningitidis B strains, after receiving a booster dose of either rMenB or rMen+OMV NZ vaccines at 40 months of age are compared with hSBA responses following one catch-up dose of rMenB+OMV NZ vaccine given at 40 months in vaccine-naive subjects.
  Baseline is defined as either the time that the (first) booster dose was given or the time of the first vaccination in this study.
Time Frame: 1 month post - booster/ -dose 1 for Naïve
Population: The analysis was done on the MITT population, booster response.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 5rMenB | 5rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 28 | 17 | 37
Percentage of subjects
  H44/76 strain | 89 [72 to 98] | 94 [71 to 100] | 41 [25 to 58]
  5/99 strain (N=27, 16, 37) | 100 [87 to 100] | 94 [70 to 100] | 68 [50 to 82]
  NZ 98/254 strain | 11 [2 to 28] | 82 [57 to 96] | 57 [39 to 73]
  M10713 strain (N=27, 15, 37) | 41 [22 to 61] | 67 [38 to 88] | 14 [5 to 29]

9. Secondary Outcome: Geometric Mean Antibody Titers in Children After Receiving Two Booster Doses of Either rMenB or rMenB+OMV NZ Vaccine at 40 & 42 Months of Age.
Description: The GMTs against N.meningitidis B strains in children (who had previously received one dose MenB vaccine in parent study) after a two booster doses of either rMenB or rMenB+OMV NZ vaccine given at 40 & 42 months of age.
Time Frame: 1 month post vaccination
Population: The analysis was done on the MITT population, booster response.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3rMenB | 3rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 13 | 8 | 38
Titers
  H44/76 strain (dose 1; N=13, 7, 38) | 94 [48 to 185] | 76 [30 to 190] | 12 [7.96 to 19]
  H44/76 strain (dose 2; N=13, 8, 36) | 127 [81 to 198] | 145 [82 to 255] | 88 [66 to 117]
  5/99 strain (dose 1; N=13, 7, 38) | 2379 [1164 to 4859] | 509 [192 to 1348] | 22 [12 to 40]
  5/99 strain (dose 2; N=13, 8, 36) | 5240 [3082 to 8911] | 2413 [1226 to 4747] | 1019 [762 to 1362]
  NZ 98/254 strain (dose 1; N=13, 7, 38) | 1.73 [0.86 to 3.48] | 148 [57 to 384] | 7.73 [4.62 to 13]
  NZ 98/254 strain (dose 2; N=13, 8, 36) | 1.86 [0.89 to 3.88] | 65 [25 to 165] | 47 [31 to 72]
  M10713 strain (dose 1; N=13, 7, 38) | 35 [18 to 68] | 30 [12 to 74] | 11 [6.7 to 19]
  M10713 strain (dose 2; N=12, 8, 36) | 21 [9.25 to 47] | 36 [13 to 98] | 33 [22 to 51]

10. Secondary Outcome: Percentage of Subjects With Serum Bactericidal Antibody Titers ≥ 1:4 and ≥ 1:8 After Receiving Two Booster Doses of Either rMenB or rMenB+OMV NZ Vaccine at 40 & 42 Months of Age.
Description: The percentages of subjects (who had previously received one dose of MenB vaccine in parent study) with hSBA ≥ 1:4 and ≥ 1:8, against N.meningitidis B strains after receiving two booster doses of either rMenB or rMenB+OMV NZ vaccine at 40 & 42 months of age.
Time Frame: 1 month post vaccination
Population: The analysis was done on the MITT population, booster response.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 3rMenB | 3rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 13 | 8 | 38
Percentages of subjects
  H44/76 strain (≥1:4 - dose 1; N=13, 7, 38) | 100 [75 to 100] | 100 [59 to 100] | 89 [75 to 97]
  H44/76 strain (≥1:4 - dose 2; N=13, 8, 36) | 100 [75 to 100] | 100 [63 to 100] | 100 [90 to 100]
  H44/76 strain (≥1:8 - dose 1; N=13, 7, 38) | 100 [75 to 100] | 100 [59 to 100] | 63 [46 to 78]
  H44/76 strain (≥1:8 - dose 2; N=13, 8, 36) | 100 [75 to 100] | 100 [63 to 100] | 100 [90 to 100]
  5/99 strain (≥1:4 - dose 1; N=13, 7, 38) | 100 [75 to 100] | 100 [59 to 100] | 76 [60 to 89]
  5/99 strain (≥1:4 - dose 2; N=13, 8, 36) | 100 [75 to 100] | 100 [63 to 100] | 100 [90 to 100]
  5/99 strain (≥1:8 - dose 1; N=13, 7, 38) | 100 [75 to 100] | 100 [59 to 100] | 71 [54 to 85]
  5/99 strain (≥1:8 - dose 2; N=13, 8, 36) | 100 [75 to 100] | 100 [63 to 100] | 100 [90 to 100]
  NZ 98/254 strain (≥1:4 - dose 1; N=13, 7, 38) | 15 [2 to 45] | 100 [59 to 100] | 66 [49 to 80]
  NZ 98/254 strain (≥1:4 - dose 2; N=13, 8, 36) | 15 [2 to 45] | 100 [63 to 100] | 94 [81 to 99]
  NZ 98/254 strain (≥1:8 - dose 1; N=13, 7, 38) | 15 [2 to 45] | 100 [59 to 100] | 58 [41 to 74]
  NZ 98/254 strain (≥1:8 - dose 2; N=13, 8, 36) | 15 [2 to 45] | 100 [63 to 100] | 94 [81 to 99]
  M10713 strain (≥1:4 - dose 1; N=13, 7, 38) | 100 [75 to 100] | 86 [42 to 100] | 76 [60 to 89]
  M10713 strain (≥1:4 - dose 2; N=12, 8, 36) | 83 [52 to 98] | 100 [63 to 100] | 89 [74 to 97]
  M10713 strain (≥1:8 - dose 1; N=13, 7, 38) | 85 [55 to 98] | 86 [42 to 100] | 61 [43 to 76]
  M10713 strain (≥1:8 - dose 2; N=12, 8, 36) | 75 [43 to 95] | 100 [63 to 100] | 86 [71 to 95]

11. Secondary Outcome: Percentage of Subjects With 4-fold Increase in Antibody Titers After Receiving Two Booster Doses of Either rMenB or rMenB+OMV NZ Vaccine at 40 & 42 Months of Age.
Description: The percentages of subjects (who had previously received one dose of MenB vaccine in parent study) displaying 4-fold increase in antibody titers over baseline against N.meningitidis B strains, after receiving two booster doses of either rMenB or rMenB+OMV NZ vaccine at 40 & 42 months of age.
Time Frame: 1 month post vaccination
Population: The analysis was done on the MITT population, booster response.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 3rMenB | 3rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 13 | 8 | 37
Percentages of subjects
  H44/76 strain (dose 1; N=13, 7, 37) | 100 [75 to 100] | 86 [42 to 100] | 41 [25 to 58]
  5/99 strain (dose 1; N=13, 7, 37) | 100 [75 to 100] | 100 [59 to 100] | 68 [50 to 82]
  NZ 98/254 strain (dose 1; N=13, 7, 37) | 15 [2 to 45] | 100 [59 to 100] | 57 [39 to 73]
  M10713 strain (dose 1; N=12, 7, 37) | 58 [28 to 85] | 57 [18 to 90] | 14 [5 to 29]
  H44/76 strain (dose 2; N=13, 8, 34) | 100 [75 to 100] | 88 [47 to 100] | 97 [85 to 100]
  5/99 strain (dose 2; N=13, 8, 34) | 100 [75 to 100] | 100 [63 to 100] | 100 [90 to 100]
  NZ 98/254 strain (dose 2; N=13, 8, 34) | 15 [2 to 45] | 100 [63 to 100] | 94 [80 to 99]
  M10713 strain (dose 2; N=11, 8, 34) | 64 [31 to 89] | 75 [35 to 97] | 53 [35 to 70]

12. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥ 1:4 and ≥1:8 Following Two Catch up Doses of rMenB+OMV NZ Vaccine Given One Month Apart, Either at 40 or 60 Months of Age.
Description: The percentage of subjects with hSBA ≥ 1:4 and ≥ 1:8 after two catch-up doses of rMenB+OMV NZ vaccine when given either at 40 & 42 months or 60 & 62 months of age are reported.
Time Frame: 1 month post -vaccine dose two
Population: The analysis was done on the MITT population, 2-dose catch-up regimen.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 36 | 42
Percentages of subjects
  hSBA ≥1:4 ( H44/76 strain) | 100 [90 to 100] | 93 [81 to 99]
  hSBA ≥1:8 (H44/76 strain) | 100 [90 to 100] | 93 [81 to 99]
  hSBA ≥1:4 (5/99 strain) | 100 [90 to 100] | 100 [92 to 100]
  hSBA ≥1:8 (5/99 strain) | 100 [90 to 100] | 100 [92 to 100]
  hSBA ≥1:4 (NZ 98/254 strain) | 94 [81 to 99] | 100 [92 to 100]
  hSBA ≥1:8 (NZ 98/254 strain) | 94 [81 to 99] | 90 [77 to 97]
  hSBA ≥1:4 (M10713 strain; N=36, 41) | 89 [74 to 97] | 100 [91 to 100]
  hSBA ≥1:8 (M10713 strain; N=36, 41) | 86 [71 to 95] | 98 [87 to 100]

13. Secondary Outcome: Geometric Mean Antibody Titers in Children After Two Catch up Doses of rMenB+OMV NZ Vaccine Given, Either at 40 or 60 Months of Age.
Description: The geometric mean antibody titers in children after two catch-up doses of rMenB+OMV NZ vaccine when given either at 40 & 42 months or 60 & 62 months of age are reported.
Time Frame: 1 month post vaccine dose two
Population: The analysis was done on the MITT population, 2-dose catch-up regimen.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 36 | 42
Titers
  H44/76 strain | 88 [63 to 123] | 34 [25 to 47]
  5/99 strain | 1019 [688 to 1510] | 865 [601 to 1244]
  NZ 98/254 strain | 47 [32 to 69] | 29 [20 to 41]
  M10713 strain (N=36, 41) | 33 [24 to 47] | 43 [31 to 59]

14. Secondary Outcome: Percentage of Subjects With a 4-fold Increase in Antibody Titers After Receiving Two Catch up Doses of rMenB+OMV NZ Vaccine, Either at 40 or 60 Months of Age.
Description: The percentages of subjects with four-fold increase in hSBA titers over baseline against N.meningitidis B one month after receiving a two catch-up doses of rMenB+OMV NZ vaccine either at 40 & 42 months or 60 & 62 months of age.
Time Frame: 1 month post vaccine dose 2
Population: The analysis was done on the MITT population, 2-dose catch-up regimen.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 34 | 38
percentage of subjects
  H44/76 strain | 97 [85 to 100] | 71 [54 to 85]
  5/99 strain | 100 [90 to 100] | 100 [91 to 100]
  NZ 98/254 strain | 94 [80 to 99] | 89 [75 to 97]
  M10713 strain | 53 [35 to 70] | 21 [10 to 37]

15. Secondary Outcome: Persisting Geometric Mean Antibody Titers Against N.Meningitidis B in Children at 60 Months of Age.
Description: The persisting GMTs against N.meningitidis B strains in children at 60 months of age who had received one or two booster doses of either rMenB or rMenB+ OMV NZ vaccine or had received two catch-up doses of rMenB+ OMV NZ vaccine at 40 months of age in the present study are compared with GMTs in vaccine-naïve subjects.
Time Frame: 18-20 months after last Men B vaccine; baseline for naïve_6062
Population: The analysis was done on the MITT, 60 months of age, antibody persistence population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 5rMenB | 5rMenB+OMV NZ | 3rMenB | 3rMenB+OMV NZ | Naive_4042 | Naive_6062
Number analyzed (Participants) | 24 | 16 | 13 | 5 | 29 | 46
Titers
  H44/76 strain (N=24, 16, 13, 5, 28, 46) | 3.13 [1.75 to 5.59] | 4.68 [2.3 to 9.52] | 18 [8.08 to 39] | 13 [3.52 to 45] | 12 [6.27 to 23] | 2.98 [1.86 to 4.78]
  5/99 strain (N=23, 16, 13, 5, 28, 46) | 43 [19 to 99] | 136 [51 to 365] | 369 [123 to 1103] | 210 [36 to 1227] | 44 [29 to 67] | 1.14 [0.88 to 1.47]
  NZ 98/254 strain | 1.05 [0.8 to 1.38] | 4.95 [3.54 to 6.92] | 1 [0.69 to 1.45] | 11 [5.93 to 20] | 2.42 [1.59 to 3.66] | 1.04 [0.96 to 1.14]
  M10713 strain (N=22, 16, 12, 5, 27, 46) | 12 [7.22 to 20] | 10 [5.67 to 19] | 12 [5.85 to 24] | 25 [8.47 to 74] | 8.52 [5.09 to 14] | 18 [12 to 28]

16. Secondary Outcome: Percentage of Subjects With Persisting Serum Bactericidal Antibodies ≥1:4 and ≥1:8 in Children at 60 Months of Age.
Description: The percentage of subjects with persisting hSBA titers ≥1:4 and ≥1:8 at 60 months of age against N.meningitidis B strains after having received one or two booster doses of either rMenB or rMenB+ OMV NZ vaccine or had received two catch-up doses of rMenB+ OMV NZ vaccine at 40 months of age in the present are reported.
Time Frame: 18-20 months after last Men B vaccine; baseline for naïve_6062
Population: The analysis was done on the MITT, 60 months of age, antibody persistence population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 5rMenB | 5rMenB+OMV NZ | 3rMenB | 3rMenB+OMV NZ | Naive_4042 | Naive_6062
Number analyzed (Participants) | 24 | 16 | 13 | 5 | 29 | 46
Percentage of subjects
  hSBA ≥1:4 (H44/76 strain; N=24, 16, 13, 5, 28, 46) | 46 [26 to 67] | 44 [20 to 70] | 85 [55 to 98] | 80 [28 to 99] | 71 [51 to 87] | 33 [20 to 48]
  hSBA ≥1:4 (5/99 strain; N=23, 16, 13, 5, 28, 46) | 83 [61 to 95] | 88 [62 to 98] | 100 [75 to 100] | 100 [48 to 100] | 100 [88 to 100] | 2 [0.055 to 12]
  hSBA ≥1:4 (NZ 98/254 strain) | 0 [0 to 14] | 69 [41 to 89] | 0 [0 to 25] | 80 [28 to 99] | 31 [15 to 51] | 2 [0.055 to 12]
  hSBA ≥1:4 (M10713 strain; N=22, 16, 12, 5, 27, 46) | 77 [55 to 92] | 88 [62 to 98] | 92 [62 to 100] | 100 [48 to 100] | 81 [62 to 94] | 83 [69 to 92]
  hSBA ≥1:8 (H44/76 strain; N=24, 16, 13, 5, 28, 46) | 25 [10 to 47] | 31 [11 to 59] | 77 [46 to 95] | 60 [15 to 95] | 61 [41 to 78] | 26 [14 to 41]
  hSBA ≥1:8 (5/99 strain; N=23, 16, 13, 5, 28, 46) | 74 [52 to 90] | 88 [62 to 98] | 100 [75 to 100] | 100 [48 to 100] | 93 [76 to 99] | 2 [0.055 to 12]
  hSBA ≥1:8 (NZ 98/254 strain) | 0 [0 to 14] | 31 [11 to 59] | 0 [0 to 25] | 40 [5 to 85] | 21 [8 to 40] | 0 [0 to 8]
  hSBA ≥1:8 (M10713 strain; N=22, 16, 12, 5, 27, 46) | 59 [36 to 79] | 63 [35 to 85] | 67 [35 to 90] | 80 [28 to 99] | 48 [29 to 68] | 70 [54 to 82]

17. Secondary Outcome: Persisting Geometric Mean Antibody Concentrations Against Vaccine Antigen 287-953 in Children (Who Had Previously Received 4 Doses of MenB Vaccine in Parent Study) at 40 Months of Age.
Description: The persisting geometric mean antibody concentrations (GMCs) against vaccine antigen 287-953 in children (at 40 months of age) who had previously received 4 doses of either rMenB or rMen+OMV NZ vaccines in parent study , are compared with the the GMCs in vaccine-naïve children.
  GMCs against vaccine antigen 287-953 were measured using enzyme linked immunosorbent assay (ELISA).
Time Frame: 28 months after last Men B vaccination; Baseline for Naïve_4042 group
Population: The analysis was done on the MITT, 40 months of age, antibody persistence population.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | 5rMenB | 5rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 28 | 17 | 38
AU/mL | 82 [59 to 113] | 62 [41 to 94] | 23 [19 to 26]

18. Secondary Outcome: Persisting Geometric Mean Antibody Concentrations Against Vaccine Antigen 287-953 in Children (Who Had Previously Received 1dose of MenB Vaccine in Parent Study) at 40 Months of Age.
Description: The persisting GMCs against vaccine antigen 287-953 in children (at 40 months of age) who had previously received 1 dose of either rMenB or rMen+OMV NZ vaccines in parent study , are compared with the the GMCs in vaccine-naïve children.
  GMCs against vaccine antigen 287-953 were measure using ELISA.
Time Frame: 28 months after last Men B vaccination; baseline for naïve_4042 group
Population: The analysis was done on the MITT, 40 months of age, antibody persistence population.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | 3rMenB | 3rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 14 | 8 | 40
AU/mL | 32 [21 to 49] | 28 [16 to 50] | 23 [19 to 26]

19. Secondary Outcome: Geometric Mean Antibody Concentrations Against Vaccine Antigen 287-953 in Children (Who Had Previously Received 4 Doses of MenB Vaccine) After Receiving One Booster Dose of Either rMenB or rMenB+OMV NZ at 40 Months of Age.
Description: The GMCs against vaccine antigen 287-953 in children (who had previously received four doses MenB vaccine in parent study) after a single booster dose of either rMenB or rMenB+OMV NZ vaccine given at 40 months of age, are compared with the GMCs following one catch-up dose rMenB+OMV NZ vaccine given at 40 months to vaccine-naive subjects.
Time Frame: 1 month post booster; 1 month post dose for naïve_4042 group
Population: The analysis was done on the MITT, 40 months of age, antibody persistence population.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | 5rMenB | 5rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 28 | 19 | 38
AU/mL | 5592 [3900 to 8017] | 3934 [2540 to 6093] | 64 [44 to 94]

20. Secondary Outcome: Geometric Mean Antibody Concentrations Against Vaccine Antigen 287-953 in Children After Receiving Two Booster Doses of Either rMenB or rMenB+OMV NZ at 40 & 42 Months of Age.
Description: The GMCs against vaccine antigen 287-953 in children (who had previously received 1 dose of either rMenB or rMen+OMV NZ vaccines in parent study) , are compared with the GMCs in children who received to catch-up doses of rMenB+OMV NZ at 40 & 42 months .
Time Frame: 1 month after each booster/ vaccine dose
Population: The analysis was done on the MITT population, booster response.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | 3rMenB | 3rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 13 | 8 | 38
AU/mL
  after 1st booster/vaccine dose (N=13, N=7, N=38) | 2100 [1100 to 4007] | 1764 [731 to 4256] | 64 [44 to 94]
  after 2nd booster/vaccine dose (N=13, N=8, N=36) | 3790 [2265 to 6342] | 3660 [1899 to 7055] | 3464 [2782 to 4313]

21. Secondary Outcome: Geometric Mean Concentrations Against Vaccine Antigen 287-953 in Children After Two Catch up Doses of rMenB+OMV NZ Vaccine Given Either at 40 or 60 Months of Age.
Description: The GMCs against vaccine antigen 287-953 in children after two catch-up doses of rMenB+OMV NZ vaccine when given either at - 40 & 42 months or 60 & 62 months of age are reported.
Time Frame: 1 month post vaccine dose two
Population: The analysis was done on the MITT population, Booster response.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 36 | 42
AU/mL | 3464 [2672 to 4489] | 1744 [1372 to 2218]

22. Secondary Outcome: Persisting Geometric Mean Concentrations Against Vaccine Antigen 287-953 in Children at 60 Months of Age.
Description: The persisting GMCs against vaccine antigen 287-953 in children at 60 months of age who had either received one or two booster doses of either rMenB or rMenB+OMV NZ vaccine or had received two catch-up doses of rMenB+OMV NZ vaccine at 40 months of age in the present are compared with GMCs in vaccine-naïve subjects.
Time Frame: 18-20 months after last Men B vaccine; baseline for naïve_6062
Population: The analysis was done on the MITT, 60 months of age, antibody persistence population population.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | 5rMenB | 5rMenB+OMV NZ | 3rMenB | 3rMenB+OMV NZ | Naive_4042 | Naive_6062
Number analyzed (Participants) | 24 | 16 | 13 | 5 | 28 | 47
AU/mL | 670 [475 to 945] | 320 [210 to 487] | 280 [175 to 447] | 250 [118 to 532] | 121 [88 to 166] | 25 [20 to 32]

23. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After a Receiving Two Catch-up Doses of rMenB+OMV NZ Vaccine Either at 40 Months or 60 Months of Age.
Description: The safety and tolerability of two catch-up doses of rMenB+OMV NZ vaccine when administered either at 40 & 42 months or 60 & 62 months of age in children is assessed in terms of number of subjects with solicited local and systemic reactions following vaccination.
Time Frame: Day 1-7 after any vaccination
Population: Analysis was done on the MITT - Two Dose Catch Up Schedule population.
Measure: Number; unit: Number of subjects
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 42 | 50
Number of subjects
  Local | 42 | 49
  Injection-site pain | 41 | 46
  Injection-site erythema | 42 | 48
  Injection-site induration | 23 | 29
  Injection-site swelling | 31 | 27
  Systemic | 38 | 42
  Changes in eating habits | 21 | 23
  Sleepiness | 25 | 23
  Vomiting | 1 | 8
  Diarrhea | 7 | 7
  Irritability | 35 | 31
  Headache | 8 | 8
  Arthralgia | 16 | 16
  Rash | 2 | 4
  Fever (≥38°C) | 7 | 6
  Other | 31 | 33
  Antipyretic preventive medication used | 30 | 33
  Antipyretic treatment medication used | 7 | 7
  Medically attended fever | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1-7 after each vaccination for Solicited AEs; Unsolicited AEs were collected throughout the study period.
Description: The analyses for the data in this section are from the safety set. Non serious AEs are reported based on MedDRA version 17.0.
Arm/Group | 5rMenB | 5rMenB+OMV NZ | 3rMenB | 3rMenB+OMV NZ | Naive_4042 | Naive_6062
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/19 | 0/14 | 0/8 | 0/42 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/19 | 0/14 | 1/8 | 2/42 | 2/50
Other Adverse Events (participants affected / at risk) | 29/29 | 19/19 | 14/14 | 8/8 | 42/42 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5rMenB (N=29) | 5rMenB+OMV NZ (N=19) | 3rMenB (N=14) | 3rMenB+OMV NZ (N=8) | Naive_4042 (N=42) | Naive_6062 (N=50)
lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
cystic lymphangioma (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5rMenB (N=29) | 5rMenB+OMV NZ (N=19) | 3rMenB (N=14) | 3rMenB+OMV NZ (N=8) | Naive_4042 (N=42) | Naive_6062 (N=50)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 3 | 1 | 8 | 7
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 3 | 0 | 1 | 8
Hyperpyrexia (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 28 | 19 | 14 | 8 | 42 | 48
Injection site induration (General disorders) | 14 | 9 | 8 | 6 | 23 | 29
Injection site pain (General disorders) | 17 | 14 | 8 | 8 | 41 | 46
Injection site swelling (General disorders) | 13 | 5 | 9 | 4 | 31 | 27
Irritability (General disorders) | 14 | 10 | 9 | 8 | 35 | 31
Local swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 7 | 0 | 7 | 6
Ear infection (Infections and infestations) | 2 | 1 | 2 | 1 | 4 | 1
Eczema infected (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 1
Nasopharingitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 2 | 0 | 4 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0
Varicella (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 6 | 4 | 4 | 16 | 16
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 8 | 8
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 13 | 12 | 8 | 6 | 25 | 23
Eating disorders (Psychiatric disorders) | 5 | 10 | 5 | 4 | 21 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 1 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days